CLINICAL TRIAL: NCT05253859
Title: CFTR Modulators and Gastrointestinal Complications
Acronym: CFTR-MAGIC
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); University of Washington (Other); Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CFTR-MAGIC
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2023-07

CONDITIONS: Cystic Fibrosis; Gastrointestinal System Disease; Distal Intestinal Obstruction Syndrome; Pancreatic Enzyme Abnormality; Pancreatic Disease; Lung Diseases; Digestive System Disease
Keywords: Cystic fibrosis; Distal Intestinal Obstruction Syndrome; Pancreatic enzyme replacement therapy; Gastrointestinal symptoms; Gut symptoms
MeSH Terms: conditions — Cystic Fibrosis; Digestive System Diseases; Pancreatic Diseases; Lung Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cystic fibrosis registry (UK): People with cystic fibrosis registered in the UK CF registry
  Interventions: Other: No intervention
- Cystic fibrosis registry (US): People with cystic fibrosis registered in the US CF registry
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Registry study: No intervention

SUMMARY:
To elucidate the similarities and distinctions in non-pulmonary manifestations of cystic fibrosis (CF) including distal intestinal obstruction syndrome (DIOS) incidence and pancreatic enzyme replacement therapy (PERT) use between US and UK CF populations in a parallel study using data from the UK and US CF registries. To assess how CFTR modulators impacted upon recorded PERT use and incidence of DIOS.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a autosomal recessive multi-system disorder caused by mutations to the cystic fibrosis transmembrane conductance regulator (CFTR) gene. As well as the documented respiratory complications of CF, gastrointestinal manifestations are of clinical importance. CFTR mutations in the gastrointestinal tract are responsible for pancreatic exocrine insufficiency in around 85% of people with CF (pwCF). In addition a severe gastrointestinal complication in CF is distal intestinal obstructive syndrome (DIOS), affecting 5.7% pwCF in the UK (2.5% in <16 years and 7.7% in adults) and 2.1% in the US (<18 years 1.7%, adult 2.4%) in 2019.

This is a parallel data registry study using data from the UK and US CF registries, with data provided for the time period 2007-2018. As such no individual participants will be recruited to the study. The CFTR modulators to be studies are Ivacaftor and lumacaftor/ivacaftor.

Study aims;

* Describe DIOS events and PERT usage in UK and US registries
* Determine the effect of CFTR modulators on the incidence of DIOS and use of PERT: population time series
* Determine the effect of CFTR modulators on the incidence of DIOS and use of PERT: patient-level time series

The outcomes of the above aims will be used to generate hypotheses regarding the effect of the newer CFTR modulators such as Symdeko/Symkevi and Tricaftor/Kaftrio on PERT usage and DIOS incidence in CF registry data post 2018. This will form the basis of future studies.

ELIGIBILITY:
Inclusion Criteria:

* All patients with CF of any genotype on the UK and US cystic fibrosis registries from the period 2007 - 2018.

Exclusion Criteria:

- Patients whose CFTR modulator status is unknown or only have one year of CFTR data recorded on the registry will be excluded from the analysis of the effects of CFTR modulators. This is to account for the fact that DIOS data is annualised on the registries, therefore there is no certainty at what time of year DIOS was diagnosed in relation to commencing CFTR modulator therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children, adolescents and adults with a diagnosis of cystic fibrosis whose data are registered on either the UK or US cystic fibrosis registries.
Sampling Method: Non-Probability Sample
Enrollment: 47023 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2024-02-10 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Describe DIOS events and PERT usage in UK and US registries 2007-2018 | 2 years
  Descriptive analysis to include cumulative incidence of DIOS and prevalence of PERT usage in the UK and US. PERT use will be dichotomised (i.e use/no use), incidence of DIOS (event/no event), plotted by year, separated by registry. Trends will be described according to age range (<6, 6-11, 12+), sex, BMI, ethnicity, antibiotic use, gastrointestinal co-morbidities and FEV1 lung function.
  These demographics will also be used for demographic propensity matching to define a control group of non-eligible non-users of CFTR modulators that are otherwise representative of the CFTR modulator user group the year that the CFTR modulator exposure was commenced.
Determine the effect of CFTR modulators on the incidence of DIOS and use of PERT: population level controlled interrupted time series (ITS) | 2 years
  This will investigate the effect of CFTR modulator intervention on the rate on PERT use and DIOS incidence.
  ITS will explore proportion of DIOS events at population level in the CFTR modulator population and the propensity score defined comparator population. ITS will explore proportion of overall PERT usage (user/non user), and the proportion of individuals with a reduction in weight standardised PERT dose (decrease/no decrease).
Determine the effect of CFTR modulators on the incidence of DIOS and use of PERT: patient-level time series | 2 years
  This will focus on patient level associations to complement the registry level findings. Associations in the incidence of PERT usage and DIOS events from 2012 in individuals taking CFTR modulators, compared to propensity matched controls will be explored.
  DIOS events: Multilevel Poisson Regression model for count data by year, incidence rate ratio (frequency of DIOS events). Adjusted analysis for main covariates.
  PERT use: Multilevel linear regression for continuous data, multilevel logistic regression for dichotomised data. Adjusted for main covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Smyth, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, United Kingdom

REFERENCES:
- See also: Original article. "Pancreatic enzyme prescription following ivacaftor licensing: A retrospective analysis of the US and UK cystic fibrosis registries" — https://doi.org/10.1016/j.jcf.2024.01.011

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/59/NCT05253859/Prot_SAP_000.pdf